CLINICAL TRIAL: NCT02086136
Title: Aortic Dissection Detection Risk Score Plus D-dimer in the Diagnostic Workup of Suspected Acute Aortic Dissection: a Prospective Multicenter Study
Brief Title: Aortic Dissection Detection Risk Score Plus D-dimer in Suspected Acute Aortic Dissection
Acronym: ADvISED
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Medical Doctor Emergency Medicine, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 1000
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Aortic Dissection
Keywords: aortic dissection; diagnosis; emergency medicine; d-dimer
MeSH Terms: conditions — Aortic Dissection; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected AD: Consecutive adult patients with suspected AD presenting to Emergency Departments will be enrolled at the time of initial medical evaluation and before the establishment of a final diagnosis.

SUMMARY:
Acute aortic dissection (AD) is a deadly, difficult to diagnose disease presenting with an array of common and unspecific symptoms. Aortic dissection detection (ADD) risk score is a bedside clinical tool to estimate the risk of AD. D-dimer has been evaluated in several studies as a biomarker of AD and has showed a pooled diagnostic sensitivity of 97%. However, considering the severe morbidity and mortality of AD, a negative d-dimer per se is considered insufficient to rule-out AD in unselected patients.

The aim of the present study is to evaluate whether the diagnostic performance of d-dimer differs in patients at different clinical risk of AD, and in particular whether a negative d-dimer test may allow safe rule-out of AD in any patient subgroup without necessity to perform urgent aortic imaging.

Consecutive adult patients with suspected AD presenting to Emergency Department will be enrolled before the establishment of a final diagnosis; a standardized clinical form comprehensive of presence/absence of 12 risk markers allowing ADD risk score fulfilled and d-dimer levels measured at presentation.

The aortic imaging exam used to confirm or refuse of AD will be computed tomography angiography or transesophageal echocardiography and final diagnosis established after reviewing of all available data.

The accuracy, failure rate and efficiency of a diagnostic strategy combining standardized clinical stratification via the ADD risk score with d-dimer testing will therefore be assessed.

DETAILED DESCRIPTION:
Acute AD will include the following etiological entities, also known as acute aortic syndromes: acute aortic dissection, intramural aortic hematoma, penetrating aortic ulcer and spontaneous aortic rupture.

A pre-specified secondary sub-analysis will evaluate the diagnostic accuracy of focus cardiac ultrasound (FoCUS) and chest x ray for suspected AD.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presentation to the ED with any of the following symptoms: chest pain, back pain, abdominal pain, syncope or symptoms of perfusion deficit (central nervous system, mesenteric, myocardial, or limb ischemia)
* Aortic dissection considered among the differential diagnosis by the attending physician. Enrollment in the study will be decided by the attending physician during evaluation in the ED and before the establishment of a final diagnosis.

Exclusion Criteria:

* An alternative diagnosis to AD objectively established by the attending physician after the initial medical evaluation
* Clinical severity or other conditions not allowing complete evaluation/proper enrollment
* Lack of consent to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients with suspected AD presenting to Emergency Departments will be enrolled at the time of initial medical evaluation and before the establishment of a final diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of ADD risk score and d-dimer in suspected aortic dissection | 2 weeks after the end of recruitment
  The diagnostic performance of d-dimer will be assessed by computing sensitivity, specificity, negative and positive predictive values and negative and positive likelihood ratios with their 95% confident interval (95% CI) in all patients and within ADD risk score classes. The ADD risk score will be calculated based on the number of categories where at least one risk marker is present. Patients will be divided in low-risk (0 risk markers, ADD risk score 0), intermediate-risk (ADD risk score 1, at least 1 risk marker in 1 ADD risk category) and high-risk (ADD risk >1, at least 1 risk marker in >1 ADD risk categories). For diagnostic accuracy analyses, also a category of non-high-risk patients (ADD risk score ≤1) will be used.

SECONDARY OUTCOMES:
Efficiency and failure rate of a diagnostic strategy using ADD risk score and d-dimer | 2 weeks after the end of recruitment
  Conventional accuracy measures, failure rate and the efficiency of d-dimer will be calculated in high-risk patients (ADD risk score >1), in low-risk patients (ADD risk score 0) and in the intermediate and low-risk patients combined (non high-risk patients, ADD risk score ≤1). Failure rate (false negative proportion) will be calculated as the number of patients with a negative d-dimer and a final diagnosis of AD divided by all patients with negative d-dimer in the same risk group. The efficiency of the diagnostic strategy will be calculated as the number of patients with a negative d-dimer within a risk group divided by all included patients.

OTHER OUTCOMES:
Secondary analysis of focus cardiac echocardiography (FoCUS) for diagnosis of aortic dissection | 2 years after after the end of recruitment
  FoCUS will be performed during the Emergency Department index visit, before conclusive diagnosis. FoCUS will assess presence/absence of the following sonographic signs: intimal flap, intramural aortic hematoma, penetrating aortic ulcer, thoracic aorta enlargement, pericardial effusion/tamponade, aortic valve regurgitation. Conventional accuracy measures of FoCUS for aortic dissection will be assessed. Also the failure rate and efficiency of diagnostic strategies integrating FoCUS with ADD risk score and d-dimer test result will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Peiman Nazerian, MD, Principal Investigator — Emergency Departmen AOU Careggi; Fulvio Morello, MD, PhD, Principal Investigator — A.O. Città della Salute e della Scienza, Molinette Hospital, Torino, Italy.
Locations (6):
- Heart Institute, University of Sao Paolo, São Paulo, Brazil
- Charitè Universitätsmedizin, Berlin, Germany
- Italy (3):
  - Emergency Department, A.O.U. Città della Salute e della Scienza di Torino, Ospedale Molinette, Turin, Piedmont
  - Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Cardiovascular Research Institute (CRIB), Basel, Switzerland

REFERENCES:
- [Derived] Nazerian P, Pivetta E, Veglia S, Cavigli E, Mueller C, de Matos Soeiro A, Leidel BA, Lupia E, Rutigliano C, Wussler D, Grifoni S, Morello F; ADvISED Investigators. Integrated Use of Conventional Chest Radiography Cannot Rule Out Acute Aortic Syndromes in Emergency Department Patients at Low Clinical Probability. Acad Emerg Med. 2019 Nov;26(11):1255-1265. doi: 10.1111/acem.13819. Epub 2019 Jul 22. PMID 31220387
- [Derived] Nazerian P, Mueller C, Soeiro AM, Leidel BA, Salvadeo SAT, Giachino F, Vanni S, Grimm K, Oliveira MT Jr, Pivetta E, Lupia E, Grifoni S, Morello F; ADvISED Investigators. Diagnostic Accuracy of the Aortic Dissection Detection Risk Score Plus D-Dimer for Acute Aortic Syndromes: The ADvISED Prospective Multicenter Study. Circulation. 2018 Jan 16;137(3):250-258. doi: 10.1161/CIRCULATIONAHA.117.029457. Epub 2017 Oct 13. PMID 29030346